CLINICAL TRIAL: NCT07318818
Title: A Phase I/II Clinical Study to Evaluate the Safety and Efficacy of P134 Cells in the Treatment of Recurrent Glioblastoma
Brief Title: A Clinical Trial of P134 Cells in Recurrent Glioblastoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSL-B2172-001
Record Dates: First submitted 2025-11-27; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Glioblastoma IDH Wildtype

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- P134 cell (Experimental)
  Interventions: Biological: P134 cell injection

INTERVENTIONS:
Biological: P134 cell injection — In this Phase 1 dose-escalation study, P134 cell dosing and safety are evaluated using an accelerated titration initial dose followed by a "3+3" design. The starting dose is 1 × 10⁸ CAR⁺ T cells, administered intratumorally or intraventricularly via an Ommaya reservoir. Three dose levels are planned:
  Level 1: 1 × 10⁸ CAR⁺ T cells, Q2W Level 2: 3 × 10⁸ CAR⁺ T cells, Q2W Level 3: 5 × 10⁸ CAR⁺ T cells, Q2W
  The dose-limiting toxicity (DLT) observation period is 28 days after the first dose for each subject.
  In Phase 2 dose expansion, one or two dose levels will be selected based on integrated safety, efficacy, and other relevant data. Each selected cohort will be expanded to 20 participants for further evaluation of safety and efficacy.

SUMMARY:
This is an open-label, single-arm, dose-escalation and expansion Phase 1/2 clinical study to evaluate the safety, tolerability and efficacy of P134 cells in the treatment of recurrent glioblastoma, to explore the MTD and RP2D, and to observe the cytokinetic profile of CAR-T cells in the cerebrospinal fluid of patients. The subjects are patients with recurrent or progressive glioblastoma who are diagnosed as grade 4 glioblastoma (IDH wild-type) by histopathology or molecular pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent.
2. 18-70 years of age (inclusive), male or female.
3. Recurrent or progressive glioblastoma, histopathologically or molecularly diagnosed consistent with grade 4 glioblastoma (IDH wild-type) (refer to WHO Classification of Central Nervous System Tumors, 5th Edition, 2021).
4. Positive CD44 or CD133 antigen expression in tumor tissue confirmed by IHC, defined as ≥1% of tumor cells showing positive CD44 or CD133 IHC staining, regardless of intensity (applicable only in Phase II dose expansion study).
5. Patient has received prior radiation therapy and/or temozolomide/bevacizumab.
6. The investigator confirmed that the patient was suitable for craniotomy cerebrospinal fluid shunt and accessory (Ommaya reservoir) implantation.

Exclusion Criteria:

1. Highly allergic constitution or history of severe allergy, or allergy to related cell products
2. Received an approved or other investigational anticancer therapy within 2 weeks prior to PBMC collection or within 5 half-lives of the agent, whichever is longer, including, but not limited to: chemotherapy, radiation therapy, surgery (except diagnostic surgery), targeted therapy, cell infusion therapy, hormone therapy (except hormone replacement therapy), and traditional Chinese medicine therapy with a clear anticancer indication (traditional Chinese medicine may undergo a 1-week washout period).
3. The adverse reactions caused by previous anti-tumor treatment have not recovered to ≤ Grade 1 as evaluated by NCI CTCAE v5.0 (except alopecia, skin pigmentation, leukoplakia, etc. which are assessed as having no safety risk).
4. Tumor metastasis to the brainstem or spinal cord.
5. Patients with primary immunodeficiency disease, autoimmune diseases requiring medication (such as Crohn 's disease, ulcerative colitis, rheumatoid arthritis, systemic lupus), or previous history of autoimmune diseases of the nervous system (such as multiple sclerosis, Parkinson' s disease).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Through study completion, an average of two and a half years
  Number of participants with treatment-related adverse events as assessed by CTCAE v6.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | Through study completion, an average of two and a half years
  Number of trial participants who achieved a complete response (CR) or partial response (PR) according to the Response Assessment in Neuro-Oncology (RANO) 2.0 criteria.

OTHER OUTCOMES:
Immunogenicity | From within 24 hours before the first CAR-T cell infusion through Day 28 after the last infusion, an average duration of five months.
  Number of patients with positive serum anti-CAR molecular antibodies
Cytokinetics | From within 24 hours before the first CAR-T cell infusion through Day 28 after the last infusion, an average duration of five months
  The number of CAR-positive (CAR+) cells in cerebrospinal fluid (CSF) measured by flow cytometry, expressed as cells per milliliter (cells/mL).

IPD SHARING:
Plan to Share IPD: No